CLINICAL TRIAL: NCT05191914
Title: Clinical Study of Fulvestrant Combined With Chidamide in the Treatment of Hormone Receptor-positive Advanced Breast Cancer Resistant to Cyclin-dependent Kinases（CDK）4/6 Inhibitors
Brief Title: Clinical Study of Fulvestrant Combined With Chidamide in the Treatment of Hormone Receptor-positive Advanced Breast Cancer Resistant to CDK4/6 Inhibitors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Tao Sun, Director, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C10
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide + fulvestrant (Experimental)
  Interventions: Drug: Chidamide+ Fulvestrant

INTERVENTIONS:
Drug: Chidamide+ Fulvestrant — Drug: Chidamide chidamide 30mg orally，Biw
  Drug: Fulvestrant Fulvestrant 500mg i.m. injections every 28 days (Cycle n Day 1) with 1 additional dose on Day 15 of Cycle 1

SUMMARY:
The trial used a multicenter, open, single-arm design in which patients were treated with Chidamide combined with Fulvestrant.The primary objective is to evaluate the preliminary efficacy and safety of Chidamide in combination with Fulvestrant.Patients included in the trial were advanced breast cancer progressing on first-line aromatase inhibitor + Cyclin-dependent kinases（CDK）4/6i rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, postmenopausal * female patients;
* histologically or cytologically confirmed hormone receptor positive (ER positive, PR positive or negative), human epidermal growth factor receptor 2 negative # breast cancer patients;
* the disease before enrollment is overall unresectable locally advanced or metastatic breast cancer, and at least one measurable lesion or no measurable lesion and bone metastasis alone patients;
* for locally advanced or metastatic breast cancer, previous progression by first-line aromatase inhibitors combined with Cyclin-dependent kinases（CDK）4/6 inhibitors;
* the total number of regimens regardless of rescue therapy or adjuvant therapy before enrollment is ≤ 3, of which the number of rescue chemotherapy regimens is ≤ 1;
* Eastern Collaborative Oncology Group（ECOG） score 0-1;
* absolute neutrophil count ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L;
* expected survival time ≥ 3 months;
* Voluntarily participate in this clinical trial and sign the written informed consent form

Exclusion Criteria:

* no measurable lesions (except simple bone metastasis), such as pleural or pericardial exudate, ascites, etc.;
* underwent major surgical procedures or significant trauma before enrollment, or patients are expected to undergo major surgical treatment;
* Patients who have previously been treated with fulvestrant or histone deacetylase inhibitors (including romidepsin, vorinostat), but have received only one cycle (≤ 2 times, d1, d15, respectively) of fulvestrant within 28 days (before enrollment) are allowed;
* known to have a history of allergy to the drug components of this protocol;
* the presence of brain (membrane) metastasis during the screening period;
* a history of immunodeficiency, including HIV test positive, or suffering from other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* uncontrolled important cardiovascular disease;
* abnormal liver function [total bilirubin > 1.5 times the upper limit of normal; alanine aminotrans（ALT）/aspartate aminotransferase（AST） > 2.5 times the upper limit of normal in patients without liver metastasis, alanine aminotrans（ALT）/aspartate aminotransferase（AST） > 5 times the upper limit of normal in patients with liver metastasis], abnormal renal function (serum creatinine > 1.5 times the upper limit of normal);
* pregnant, lactating female patients or women of childbearing potential baseline pregnancy test positive; or during the study and the last dose of at least 8 to take effective contraceptive measures in subjects of childbearing age;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study (such as: severe hypertension, diabetes, thyroid disease, active infection, etc.);
* History of definite neurological or psychiatric disorders, including epilepsy or dementia;
* Unsuitable for participation in the study as judged by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-07 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 16 months
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 16 months
  Overall response rate (ORR) is defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.
Overall Survival (OS) | Up to approximately 38 months
  Time from date of randomization to the date of death from any cause.
Clinical Benefit Rate (CBR) | Up to approximately 16 months
  Clinical benefit rate (CBR), defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1.
Duration of Response (DOR) | Up to approximately 16 months
  Time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer as defined in RECIST 1.1.